CLINICAL TRIAL: NCT04007783
Title: Validation of the O-bridge Protocol, Ensuring Immediate or Delayed Prosthetic Rehabilitation in Oncology Patients Undergoing Jaw Reconstruction: a Prospective, Multicenter Trial
Brief Title: Validation of the O-bridge Protocol: a Prospective, Multicenter Trial
Status: Recruiting | Type: Observational
Sponsor: AZ Sint-Jan AV (Other)
Responsible Party: Principal Investigator, Johan Abeloos, head of department, AZ Sint-Jan AV
Other Study IDs: B322201731284
Record Dates: First submitted 2019-02-13; First posted 2019-07-05 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Benign or Malignant Tumour of the Oral Cavity; Stage III-IV Osteonecrosis; Mandibular Reconstruction; Fixed Dental Restoration; Quality of Life

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Surgical reconstruction to restore oral function and aesthetics after major ablative surgery in the oral cavity forms a challenge to maxillofacial surgeons, and greatly impacts patient' quality of life (QOL). The "Oncological-bridge (O-bridge®)" protocol, which offers (immediate/delayed) fixed prosthetic rehabilitation in a minimum of sessions and a strongly reduced two-week treatment time.

DETAILED DESCRIPTION:
Surgical reconstruction to restore oral function and aesthetics after major ablative surgery in the oral cavity forms a challenge to maxillofacial surgeons, and greatly impacts patient' quality of life (QOL). The "Oncological-bridge (O-bridge®)" protocol, which offers (immediate/delayed) fixed prosthetic rehabilitation in a minimum of sessions and a strongly reduced two-week treatment time.

Objective: The investigators aim to demonstrate the added value of the "O-bridge® protocol" in a larger sample size of at least 20 patients eligible for (immediate/delayed) fixed prosthodontic rehabilitation at time of oral cavity (mandibular) reconstruction study design: a prospective, observational cohort study. The "O-bridge® protocol", in which the standardized concept of implant loading and that of oral cavity (mandibular) reconstruction are combined with an adapted prosthetic manufacturing protocol, will be offered to eligible patients requiring ablative surgery because of a benign or malignant tumour of the oral cavity or stage 3-4 osteonecrosis.

All patients will be screened by the local maxillofacial surgeon and the prosthodontist to determine eligibility for the procedure. Imaging will be performed as part of routine surgical preparation. Clinical function, as measured with the 11-item scale by Rogers and intelligibility of speech will be assessed by the speech therapist and/or appointed health care employee prior to surgery, 3 months post-surgery and/or at time of implant placement, and at 6 weeks after placement of the O-bridge®. In addition, EORTC quality of life C30 and HN35 questionnaires will also be completed at those time-points, and at 6 months after placement of the O-bridge®. Speech-, food- and prosthetic fit-related items from the Oral Health Impact Profile (OHIP) questionnaire will be completed at 6 weeks and at 6 months after placement of the O-bridge®. Parameters related to implant and bridge stability and patient satisfaction, measured through a 10-point visual analogue scale, will be assessed at 6, 12, 24, 36, 48 and 60 months at routine follow-up consultation after placement of the O-bridge®.

As a primary endpoint, the investigators aim to demonstrate that the O-bridge® protocol significantly improves short-term patient' quality of life.

Moreover, the investigators aim to demonstrate the validity and reliability of the O-bridge® protocol, based on its short- and long-term biologic implant stability and mechanical stability of the prosthesis. In addition, they aim to measure the impact of the O-bridge® on speech intelligibility.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a histologically or clinically confirmed diagnosis of ORN, MRONJ, as classified by respectively Lyons et al. (Lyons, et al., 2014) and Ruggiero et al. (Ruggiero, et al., 2009) (Ruggiero, et al., 2014) or a benign or malignant tumour located in the oral cavity and jaw bone (NCCN, 2015) (Sobin, et al., 2009), requiring marginal, segmental or total jaw resection
* Patients eligible for jaw and oral cavity reconstruction combined with immediate/delayed implant loading for fixed prosthetic rehabilitation
* Patients not eligible for conventional removable prosthetic rehabilitation

Exclusion Criteria:

* Patients not eligible to the abovementioned criteria
* Patients with a clinically confirmed diagnosis of osteonecrosis not related to an oncological diagnosis or treatment
* Patients with medical contraindications for jaw reconstruction combined with immediate implant loading for fixed prosthetic rehabilitation
* Patients whose maternal language is non-Dutch or non-English will be excluded from the acoustic speech evaluation. A perceptual evaluation of speech intelligibility can still be performed.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: ORN, MRONJ, benign or malignant tumour in the head and neck region requiring ablative oral cavity resection including marginal, segmental or total bony jaw resection
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2017-03-04 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
EORTC QLQ C30, for measurement of quality of life | 6 weeks after O-bridge placement
  short-term quality of life after dental restoration with the O-bridge, measured through the EORTC QLQ C30 questionnaire
EORTC QLQ H&N35, for measurement of quality of life | 6 weeks after O-bridge placement
  short-term quality of life after dental restoration with the O-bridge, measured through the EORTC QLQ HN35 questionnaire
EORTC QLQ C30, for measurement of quality of life | 6 months after O-bridge placement
  short-term quality of life after dental restoration with the O-bridge, measured through the EORTC QLQ C30
EORTC QLQ H&N35, for measurement of quality of life | 6 months after O-bridge placement
  short-term quality of life after dental restoration with the O-bridge, measured through the EORTC QLQ HN35
OHIP, for measurement of quality of life | 6 weeks after O-bridge placement
  short-term quality of life after dental restoration with the O-bridge, measured through the OHIP questionnaire
OHIP, for measurement of quality of life | 6 months after O-bridge placement
  short-term quality of life after dental restoration with the O-bridge, measured through the OHIP questionnaire

SECONDARY OUTCOMES:
percentage of patients with marginal bone loss around implants | until one year post implantation
  short-term biologic implant stability, measured through OPG imaging
percentage of patients with marginal bone loss around implants | until five years post implantation
  long-term biologic implant stability, measured through OPG imaging
percentage of patients with mechanical stability problems of the prosthesis | until one year post implantation
  short-term, measured through clinical evaluation
percentage of patients with mechanical stability problems of the prosthesis | until five years post implantation
  long-term, measured through clinical evaluation
percentage of patients with difficulties in speech intelligibility | prior to and 6 weeks post O-bridge
  impact of the O-bridge on speech intelligiblity, measured through reading of a predefined oronasal text interpreted by the speech and language pathologist

CONTACTS AND LOCATIONS:
Overall Officials: Johan Abeloos, MD, Principal Investigator — AZ Sint-Lucas Brugge
Locations (5):
- Belgium (5):
  - Ziekenhuis Netwerk Antwerpen, Antwerp
  - ZMACK association - Antwerp University Hospital, Antwerp
  - Division of Oral and Maxillofacial Surgery, Department of Surgery, AZ Sint-Jan Brugge-Oostende AV, Bruges
  - University Hospital Leuven, Leuven
  - AZ Nikolaas, Sint-Niklaas

IPD SHARING:
Plan to Share IPD: No